CLINICAL TRIAL: NCT00215956
Title: A Phase I Study of Oral Topotecan as a Radiosensitizing Agent in Patients With Rectal Carcinoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-12349; USFIRB#5881
Record Dates: First submitted 2005-09-19; First posted 2005-09-22 (Estimated); Last update posted 2013-12-23 (Estimated); Status verified 2009-01

CONDITIONS: Rectal Neoplasms
Keywords: Topotecan; Rectal Neoplasms; Radiosensitizing
MeSH Terms: conditions — Rectal Neoplasms | interventions — Topotecan; Radiation; Surgical Procedures, Operative

ARMS (1):
- Dose Escalation and Radiation, Followed by Surgery (Experimental): Preoperative treatment with radiation and oral topotecan for up to 5 weeks, followed by surgery.
  Interventions: Drug: topotecan; Procedure: radiation; Procedure: surgery

INTERVENTIONS:
Drug: topotecan — Preoperative treatment: oral topotecan 5 days per week for up to 5 weeks
Procedure: radiation — Preoperative radiation
Procedure: surgery — surgery to remove tumor 4 to 8 weeks following completion of preoperative treatment

SUMMARY:
This is an open-label, single center, phase I study designed to determine the MTD or oral topotecan as a radiosensitizing agent in the treatment of rectal cancer patients. Sequential cohorts of three patients will be given increasing doses of oral topotecan and fixed doses of concurrent radiation (45GY) over five weeks.

DETAILED DESCRIPTION:
This is an open-label, single center, phase I study designed to determine the MTD or oral topotecan as a radiosensitizing agent in the treatment of rectal cancer patients. Sequential cohorts of three patients will be given increasing doses of oral topotecan and fixed doses of concurrent radiation (45GY) over five weeks. The starting dose of oral topotecan is 0.25mg/m2 to be concomitantly administered with radiation (45Gy) x 5 days every week unless the radiation is interrupted for Holidays/Weekends or toxicity requiring treatment delays occurs.

A total of 25 doses is planned. Doses will be escalated in 0.15 mg/m2 increments thereafter in subsequent cohorts. Topotecan will be administered immediately before daily radiation.

All patients will undergo a rectal biopsy before treatment begins and during treatment. Tissue will be submitted to H. Lee Moffitt Cancer Center for tumor marker assays. Tissue from the excised tumor at the time of surgery will also be sent for the same studies. Between day 10 and 14 of treatment, colonoscopy/sigmoidoscopy is mandatory to ensure having a quantitative estimate of the tumor shrinkage and to obtain a repeat rectal biopsy. All patients will undergo radiation therapy concurrently with oral topotecan. Patients will receive 180 cGY per fraction to a total dose of 4500cGy(conventional fractionation) to the pelvis using a 3 or 4 filed technique and high energy photons. Standardized fields for rectal cancer will be used to include the true pelvis (mid sacrum to at least 2-3 centimeters below the inferior aspect of the tumor volume).

Patients will undergo surgery-either a low anterior resection, abdominoperineal resection or local excision. All patients will be offered postoperative adjuvant chemotherapy consisting of 5-Fluorouracil (F-FU) 350 mg/m2/day i.v. for 5 days administered every 28 days times four cycles. Immediately prior to the administration of 5-FU, leucovorin will be administered at a dose of 20 mg/m2/day i.v. push daily for 5 days every 28 days times four cycles.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically confirmed rectal cancer.
* Written Informed Consent
* Patients should be a candidate for preoperative radiotherapy
* A primary tumor of 3cm or greater with a clinical stage of T2, T3 or T4 and any N according to the Astler-Coller modification of the Dukes staging system
* Patient must be 18 years of age or older
* Must have an ECOG performance status of 2 or Less
* Diagnosis of rectal cancer should be no more than 90 days from initial clinic visit or from the start of therapy
* Patients must be seen and evaluated at the H. Lee Moffitt Cancer Center
* Patients must be recovered from prior surgery
* Patients must have a life expectancy of 3 months or greater
* Laboratory criteria: WBC of 3,500/mm3 or greater; Neutrophils of 1,500mm3 or greater; Platelet count of 100,000/mm3 or greater; Serum creatinine of 1.5 mg/dl or lesser; or creatinine clearance of greater than 60ml/min; SGOT/AST & SGPT/ALT & alkaline phosphatase of 2 times or lesser than the upper limit or normal if liver metastases are present; Serum bilirubin of 1.5mg/dl or lesser.

Exclusion Criteria:

* Patients with their primary tumor totally excised at time of diagnosis
* Patients with recurrent rectal cancer that failed initial treatment
* Patients previously treated with topotecan
* Patients with active infection
* Any known primary or secondary immunodeficiencies
* Any condition of the GI tract which would affect GI absorption or motility (e.g., autonomic neuropathy, active gastric or duodenal ulcers or certain gastrointestinal surgeries). Patients receiving medication to maintain motility or gastric emptying are also excluded.
* Patients with uncontrolled emesis, regardless of etiology.
* Concomitant malignancies or previous malignancies within the last five years, with the exception of adequately treated basal or squamous cell carcinoma of the skin, carcinoma in situ of the cervix or a low grade prostate cancer.
* Concurrent severe medical problems unrelated to the malignancy which would significantly limit full compliance with the study or expose the patient to significant risk.
* Patients of child bearing potential, not practicing adequate contraception (barrier method or IUD for three months before the start of the study an agree to continue for at least 4 weeks after the end of the study)
* Patients who are pregnant or lactating
* Use of an investigational drug within 30 days or 5 half-lives (whichever is longer) preceding the first dose of study medication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2001-11; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of Topotecan | up to 5 weeks
  Dose escalation to determine MTD that can be given with radiation.
Side Effect Profile of Topotecan | Up to 5 weeks
  Review of adverse events

SECONDARY OUTCOMES:
Response Rate | Up to 12 weeks
  To determine pathologic response to treatment and assessment of sphincter preservation.

CONTACTS AND LOCATIONS:
Overall Officials: William Dinwoodie, MD, Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center & Research Institute, Tampa, Florida, United States